CLINICAL TRIAL: NCT01320501
Title: Real Life Experience of Erlotinib in Patients With Advanced Non-Small Cell Lung Cancer in the Middle Eastern Countries (REALME)
Brief Title: Experience of Erlotinib in Patients With Advanced Non-Small Cell Lung Cancer
Acronym: REALME
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in enrolling patients
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC08/29
Record Dates: First submitted 2011-03-19; First posted 2011-03-22 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erlotinib (Experimental): 150 mg PO daily
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — All patients will receive: TarcevaTM 150mg/day PO.

SUMMARY:
An open-label, prospective, single-arm, multi-center phase IV clinical trial of TarcevaTM as single agent

DETAILED DESCRIPTION:
Advanced NSCLC remains largely fatal, with the positive impact of chemotherapy limited by intrinsic and acquired resistance, manifested clinically by early progression and transient responses. Current chemotherapy regimens have limited efficacy with a magnitude of survival benefit that is still modest, and lead to significant toxicity, with many patients unable to receive this kind of treatment, even in first line setting. There is, therefore, a great need to provide patients with less toxic agents such as the novel targeted therapies, with the potential to improve the efficacy and maintain a good quality of life with little associated toxicity. TarcevaTM has shown benefit as single agent in pretreated patients who have progressed despite platinum-based chemotherapy as summarized in section 1.2 with minimal toxicity compared to chemotherapy, and also is currently assessed as first line treatment in advanced NSCLC with promising preliminary efficacy results.

As previously described, TarcevaTM has recently been shown to prolong survival in a large, randomized, placebo-controlled Phase III trial including 731 NSCLC patients no longer candidates for further chemotherapy. This is the first and so far the only evidence of definitive clinical benefit provided by an EGFR inhibitor in cancer patients. TarcevaTM is the standard of care for second and third line treatment for lung cancer in USA and Europe. However, the experience with this agent in the Middle Eastern population is very limited. The rationale for this program is to evaluate the pattern of TarcevaTM use in patients with advanced (inoperable stage III or IV) NSCLC who have failed standard treatment, or patients who can not receive other systemic anticancer therapy, or patients who are not medically suitable for chemotherapy (e.g., poor performance status). This will also enable us to study the efficacy and safety of TarcevaTM in this population, as there may be differences in the pharmacogenomic of this population and the previously studied population.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological documented diagnosis of inoperable, locally advanced, recurrent or metastatic (Stage IIIB or Stage IV) NSCLC.
2. Patients must have evidence of disease but measurable disease is not mandatory.
3. 18 years of age or older.
4. ECOG performance status of 0 - 3.
5. Life expectancy of at least 12 weeks.
6. Patients who received one or two previous line of systemic chemotherapy irrespective of EGFR mutation status.
7. No more than 2 prior chemotherapy regimens are permissible. Patients must have recovered from any toxic effects and at least 3-4 weeks must have elapsed from the last dose and prior to registration (14 days for vinorelbine or other vinca alkaloids or gemcitabine). Patients who, in the opinion of the investigator, have fully recovered from surgery in less than 4 weeks may also be considered for the study. Patients must have recovered (CTC < 1) from acute toxicities of any previous therapy.
8. Patients are eligible to receive Erlotinib (TarcevaTM) as first line if they met one of the following criteria:

   1. Positive EGFR mutation tested in certified lab (although EGFR test is not mandatory only if available).
   2. Poor performance status of 3
   3. Severe co morbidities and illness which make the patient not candidate for standard systemic chemotherapy .
9. .Patient with negative EGFR mutation are still candidate for 2nd and 3rd line therapy (although EGFR test is not mandatory only if available).
10. Prior radiotherapy is allowed.
11. Granulocyte count > 1.5 x 109/L and platelet count > 100 x 109/L.
12. Serum bilirubin must be < 1.5 upper limit of normal (ULN).
13. AST and ALT < 2 x ULN (or < 5 x ULN if clearly attributable to liver metastasis).
14. Serum creatinine < 1.5 ULN or creatinine clearance > 60 ml/min.
15. Able to comply with study and follow-up procedures.
16. For all females of childbearing potential a negative pregnancy test must be obtained within 72 hours before starting therapy. Patients with reproductive potential must use effective contraception.
17. Signed Informed Consent to participate in the study.

Exclusion Criteria:

1. Any unstable systemic disease (including active infection, grade 4 hypertension, unstable angina, congestive heart failure, hepatic, renal or metabolic disease).
2. Prior therapy with systemic anti-tumor therapy with HER1/EGFR inhibitors (as small molecule or monoclonal antibody therapy).
3. Any other malignancies within 5 years (except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer).
4. Patients are excluded if they have brain metastasis or spinal cord compression that is newly diagnosed and/or has not yet been definitively treated with surgery and/or radiation; previously diagnosed and treated CNS metastases or spinal cord compression with evidence of stable disease (clinically stable imaging) for at least 2 months is permitted.
5. Any significant ophthalmologic abnormality, especially severe dry eye syndrome, keratoconjunctivitis sicca, Sjogren syndrome, severe exposure keratitis or any other disorder likely to increase the risk of corneal epithelial lesions. The use of contact lenses is not recommended during the study. The decision to continue to wear contact lenses should be discussed with the patient's treating Oncologist and the ophthalmologist.
6. Patients who cannot take oral medication, who require intravenous alimentation, have had prior surgical procedures affecting absorption, or have active peptic ulcer disease.
7. Nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the pattern of use of TarcevaTM in Middle Eastern patients with advanced NSCLC | 3 years

SECONDARY OUTCOMES:
To evaluate the activity and tolerability of TarcevaTM in this patient population | 3 years
  To evaluate the activity and tolerability of TarcevaTM in this patient population, assessing:
  * Best response (as per investigator's assessment).
  * Progression-Free Survival (PFS).
  * Overall Survival (OS).
  * Safety (Serious Adverse Events (SAEs), AEs leading to premature withdrawal, unexpected and expected TarcevaTM related AEs).
  * To assess the degree of association (correlation) of EGFR expression rate (HER1) and other markers potentially predictive for response.

CONTACTS AND LOCATIONS:
Overall Officials: Abdulrahman Jazieh, MD/MPH, Principal Investigator — King Abdul Aziz Medical City for National Guard
Locations (1):
- King Abdul Aziz Medical City for National Guard Health Affairs, Riyadh, Saudi Arabia